CLINICAL TRIAL: NCT01906580
Title: Combination or Sequential Therapy of Peginterferon Alfa-2a and Entecavir for Hepatitis B e Antigen-positive Patients With Chronic Hepatitis B
Brief Title: Combination or Sequential Therapy of Peginterferon Alfa-2a and Entecavir for Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011030D
Record Dates: First submitted 2013-05-30; First posted 2013-07-24 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Hepatitis B
Keywords: HBV; entecavir; peginterferon
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peg-IFNα-2a monotherapy (Experimental): Participants will receive 180ug peg-IFNα-2a therapy for 72 weeks, and then followed to 96 weeks.
  Interventions: Drug: Peg-IFNα-2a
- Sequential therapy (Experimental): Participants will receive entecavir monotherapy for 12 weeks, and 180ug peg-IFNα-2a therapy is added for the following 12 weeks. After that, entecavir will be stopped and 180ug peg-IFNα-2a monotherapy for the following 48 weeks. All participants will followed to 96 weeks.
  Interventions: Drug: Peg-IFNα-2a; Drug: Entecavir
- Combination therapy (Experimental): Participants will receive 180ug peg-IFNα-2a combined with entecavir therapy for 72 weeks, and then followed to 96 weeks.
  Interventions: Drug: Peg-IFNα-2a; Drug: Entecavir

INTERVENTIONS:
Drug: Peg-IFNα-2a — 180ug peg-IFNα-2a, subcutaneous injection per week
  Other Names: peginterferon alfa-2a
Drug: Entecavir — 0.5mg,oral administration every day
  Other Names: Baraclude
  Arms: Combination therapy; Sequential therapy

SUMMARY:
Currently, seven medications are approved for the treatment of hepatitis B: two formulations of interferon and five nucleons(t)ide analogues. The current treatment strategy of chronic hepatitis B is now standard: initial selection of entecavir, tenofovir, or peginterferon alfa-2a (peg-IFNα-2a). Interferon is administered for a finite duration while nucleotide analogues are usually administered for many years. But among hepatitis B e antigen （HBeAg） positive patients with high serum hepatitis B virus DNA levels, the rates of virological response are poor. And antiviral drug resistance is a major limiting factor to the success of nucleotide analogue treatment. Therefore, combination therapy using peginterferon with an oral agent with a high genetic barrier to resistance might be superior to standard current monotherapy. However, the addition of lamivudine to peg-IFNα-2a therapy led to a greater decrease in serum HBV DNA levels during treatment but did not increase the rate of HBeAg sero¬conversion. Entecavir is a nucleoside analogue superior to lamivudine and adefovir in achieving higher virological response, histological improvement and normalisation of ALT. Moreover, Entecavir has a high genetic barrier with a very low incidence of drug resistance. This study is aimed to investigate the efficacy of combination or sequential therapy using peg-IFNα-2a and entecavir in HBeAg-positive chronic hepatitis B(CHB) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥16 years
2. HBsAg positive for more than 6 months, and HBeAg detection is positive for two times in 6 months before enrollment
3. Serum HBVDNA >2×10^4IU/ml
4. 80U/L < serum ALT < 400U/L, and TBIL < 34 umol/L
5. Serum ALT < 80U/L, but hepatic inflammation scores ≥ G2 or hepatic fibrosis stage ≥ S3

Exclusion Criteria:

1. Co-infected with HCV, HDV or HIV, or autoimmune liver diseases combined
2. Hepatic decompensation
3. received antiviral therapy or immunosuppressant drugs before 6 months prior to enrollment
4. Blood routine examination: WBC <3×10^9/L，neutrophile granulocyte < 1.5×10^9/L，PLT <80×10^9/L
5. Renal function: creatinine >1.5 times of upper normal limit
6. Alcoholism or a history of addiction and abuse
7. Combined with hepatocarcinoma

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
the rates of HBeAg seroconversion | at week 72

SECONDARY OUTCOMES:
normalisation of ALT | at week 2、4、12、24、36、48、60、72、84、96
liver histological improvement | at baseline and at week 72
The rates of HBsAg negative | at week12、24、36、48、60、72、84、96
the rate of virological response | at week 4、12、24、36、48、60、72、84、96
the rate of HBeAg negative | at week 12、24、36、48、60、72、84、96

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Research Center for Biological Therapy, The Institute of Translational Hepatology, Beijing 302 Hospital, Beijing, China

REFERENCES:
- [Background] Kwon H, Lok AS. Hepatitis B therapy. Nat Rev Gastroenterol Hepatol. 2011 May;8(5):275-84. doi: 10.1038/nrgastro.2011.33. Epub 2011 Mar 22. PMID 21423260
- [Background] Ayoub WS, Keeffe EB. Review article: current antiviral therapy of chronic hepatitis B. Aliment Pharmacol Ther. 2011 Nov;34(10):1145-58. doi: 10.1111/j.1365-2036.2011.04869.x. Epub 2011 Oct 7. PMID 21978243
- [Background] Kuo A, Gish R. Chronic hepatitis B infection. Clin Liver Dis. 2012 May;16(2):347-69. doi: 10.1016/j.cld.2012.03.003. PMID 22541703
- [Background] Rehermann B, Nascimbeni M. Immunology of hepatitis B virus and hepatitis C virus infection. Nat Rev Immunol. 2005 Mar;5(3):215-29. doi: 10.1038/nri1573. PMID 15738952